CLINICAL TRIAL: NCT04564729
Title: Shared Decision Aid for Post-Total Knee Arthroplasty Opioid Prescribing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Naida Margaret Cole, Anesthesiologist, University of Chicago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P002342
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Knee Arthroplasty, Total; Analgesia; Opioid Use, Unspecified
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Masking Description: Investigators not involved in administering the SDA and data collection will be blinded. The study subject and investigator(s) involved in administering the SDA and collecting outcomes data will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid (Experimental): The shared decision aid (SDA) includes factual information about the World Health Organization pain ladder, the 0-10 numeric rating score pain scale, pharmacologic pain management options, opioid medication benefits and risks and predicted post-discharge opioid requirements based on previous modeling in total knee arthroplasty patients. Subjects in the decision aid group will view the decision aid and have the opportunity to participate in shared decision-making for their discharge opioid prescriptions.
  Interventions: Other: Shared Decision Making
- Control (No Intervention): Subjects in the control group will undergo standard care and discharge practices. Baseline pain and psychosocial factors will be documented as well as postoperative pain and analgesic consumption.

INTERVENTIONS:
Other: Shared Decision Making — The intervention group will receive a shared decision-making intervention including a decision aid and conversation with a study investigator. The intervention group will have the opportunity to choose the number of opioid pills they receive at discharge from hospital after total knee arthroplasty.
  Arms: Decision Aid

SUMMARY:
This will be a randomized controlled clinical trial in patients who have undergone primary unilateral total knee arthroplasty at Brigham and Women's Faulkner Hospital, Brigham and Women's Hospital and University of Chicago Medical Center. Study subjects will receive either a shared decision aid (SDA) about pain management or standard of care at the time of discharge. The impact of the SDA on the number of leftover opioid pills on postoperative day 30 and average NRS pain score on postoperative day 7 will be assessed.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial for primary, unilateral total knee arthroplasty (TKA) patients at Brigham and Women's Faulkner Hospital, Brigham and Women's Hospital and University of Chicago Medical Center to determine the impact of using a SDA on the number of leftover opioid pills on postoperative day 30 and average NRS pain score on postoperative day 7.

The SDA includes factual information about the World Health Organization pain ladder, the 0-10 NRS pain scale, pharmacologic pain management options, opioid medication benefits and risks and predicted post-discharge opioid requirements based on previous modeling in TKA patients. The SDA has been developed by the principal investigator solely for the purpose of this study.

Patients will be enrolled on postoperative day 0 or 1 and randomized to intervention or control groups. The intervention group will view the SDA slides on the study iPad. SDA viewing will be guided by the research assistant, who will read a pre-written script as each slide is viewed. Following the guided viewing of the SDA, subjects in the intervention group will have the opportunity to ask questions to the research assistant to confirm their comprehension of the presented facts. The control group will receive no intervention and will receive standard of care and standard discharge prescriptions. The intervention group subjects will choose the number of opioid pills they wish to include in their discharge opioid prescription (anywhere from 0 to the maximum allowable as determined by clinical practice and/or state law).

Daily analgesic intake, adverse effects and numeric rating scale (NRS) pain scores will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral TKA under spinal anesthesia at Brigham & Women's Faulkner Hospital (BWFH), Brigham and Women's Hospital or University of Chicago Medical Center by a participating surgeon
* >18 years of age
* Planned discharge with the typical analgesic medications prescribed at discharge:

  * standing around-the clock Tylenol with or without an NSAID
  * tramadol PRN
  * hydromorphone (dilaudid) or oxycodone PRN

Exclusion Criteria:

* Diagnosis of dementia
* <18 years old
* Contraindication or allergy to opioids
* Contraindication or allergy to Tylenol
* Contraindication or allergy to gabapentin
* History of substance use disorder
* Preoperative pain requiring a >1-month prescription for >/=45 daily MMEs
* 4 or more preoperative analgesic prescriptions
* Hospital admission >1 day
* Discharge to a skilled nursing facility/inpatient rehabilitation center
* Non-English speaking patients
* Requirement for general anesthesia intra-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Leftover opioid pills | 30 days postoperatively
Average 0-10 NRS pain score | postoperative day 7

SECONDARY OUTCOMES:
Quantity of opioid consumed | 30 days postoperatively
Satisfaction with pain management | 30 days postoperatively
Quantity of opioid pills prescribed | postoperative day 1 at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Naida Cole, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No